CLINICAL TRIAL: NCT05533255
Title: Clinical Evaluation of Preheated Resin Composites Compared With Conventional Resin Composites in the Treatment of Noncarious Cervical Lesions - A Randomised Controlled Trial
Brief Title: Preheated Composites Vs. Conventional Composites in Noncarious Cervical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manipal University College Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Anchu Rachel Thomas, Associate Professor Dr., Manipal University College Malaysia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MUCM/FOD/AR/B10/E C-2022 (04)
Record Dates: First submitted 2022-07-16; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Noncarious Cervical Lesions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preheated Resin Composites (Experimental): Preheated resin composite is placed on the noncarious cervical lesion of a canine/ first premolar/ second premolar/ first molar on either one quadrant of the maxillary arch.
  Interventions: Other: Preheated composite resin (3M™ Filtek™ Z350 XT Universal Restorative)
- Conventional Resin Composites (Active Comparator): Conventional resin composite is placed on the noncarious cervical lesion of a canine/ first premolar/ second premolar/ first molar on the other quadrant of the maxillary arch.
  Interventions: Other: Conventional composite resin (3M™ Filtek™ Z350 XT Universal Restorative)

INTERVENTIONS:
Other: Conventional composite resin (3M™ Filtek™ Z350 XT Universal Restorative) — Composite resin at room temperature is used.
  Arms: Conventional Resin Composites
Other: Preheated composite resin (3M™ Filtek™ Z350 XT Universal Restorative) — Conventional composite resin (3M™ Filtek™ Z350 XT Universal Restorative) is preheated to a temperature of 57 degrees Celsius using a composite warmer for 10 minutes is used.
  Arms: Preheated Resin Composites

SUMMARY:
Preheating resin composites is the warming of resin composites by using a heating device (composite warmer) before its placement. Preheating increases the flow properties and allows better adaptation to cavity preparation. The high thermal energy also improves polymerization rate, thereby reducing microleakage. Conventional composites resin is used as one-paste light-cured systems, which are built up in increments to overcome the effects of setting shrinkage and to ensure thorough curing.

Several studies report failure of cervical restorations of noncarious cervical lesions and an incessant search for the most suitable restorative material. Therefore, this study aims to evaluate the clinical performance of conventional resin composites compared with preheated resin composites in the treatment of noncarious cervical lesions. Our null hypothesis states that there is no difference between the clinical performance of preheated resin composites and conventional resin composites in the treatment of noncarious cervical lesions.

This study will be conducted at the Conservative and Endodontics Department in Polyclinic B, Faculty of Dentistry, Manipal University College Malaysia (MUCM). It involves forty-six randomly selected patients with two similar noncarious cervical lesions, each on a canine, first premolar, second premolar or first molar on the contralateral side of the maxillary arch. One lesion will be restored with preheated resin composite (3M™ Filtek™ Z350 XT Universal Restorative) while the other lesion will be restored with conventional resin composite (3M™ Filtek™ Z350 XT Universal Restorative). Both restorations will be done on each patient's first visit. The patients will be recalled 1,3 and 6 months later for assessment of the restorations, using modified US Public Health Service (USPHS) criteria: marginal integrity, marginal discoloration, wear, retention, secondary caries and postoperative sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are systemically healthy (ASA I and ASA II )44 and have satisfactory oral hygiene (OHI-S score of 0 to 3.0).
* Participants must have two noncarious cervical lesions (abrasion/abfraction), each on a canine, 1st premolar, 2nd premolar or 1st molar on the contralateral side of same dental arch (maxillary arch) with similar depth and width.
* Both NCCLs are in contact with antagonist teeth as well.

Exclusion Criteria:

* Participants requiring dental prostheses of the target teeth.
* Participants have a diagnosis of caries coincident with the cervical lesion, or an indication for irreversible endodontic treatment of the target teeth.
* Existence of periodontal damage with respect to the target teeth.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Evaluation of Preheated Resin Composite Compared with Conventional Resin Composite | 1 month
  The restorations are evaluated using the modified US Public Health Service (USPHS) criteria
Clinical Evaluation of Preheated Resin Composite Compared with Conventional Resin Composite | 3 month
  The restorations are evaluated using the modified US Public Health Service (USPHS) criteria
Clinical Evaluation of Preheated Resin Composite Compared with Conventional Resin Composite | 6 month
  The restorations are evaluated using the modified US Public Health Service (USPHS) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sy Ying Heng, Principal Investigator — Manipal University College Malaysia; Sze Yee Tan, Principal Investigator — Manipal University College Malaysia; Chi Rou Tee, Principal Investigator — Manipal University College Malaysia; Krystell Chiu Yan Lau, Principal Investigator — Manipal University College Malaysia
Locations (1):
- Manipal University College Malaysia, Malacca, Malaysia

IPD SHARING:
Plan to Share IPD: No